CLINICAL TRIAL: NCT02629445
Title: High Frequency Low Energy Pacing to Terminate Fast Ventricular Arrythmias
Brief Title: HIPACE High Frequency Low Energy Pacing to Terminate Fast Ventricular Arrythmias
Acronym: HIPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CD14/11241
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cardiac Resynchronisation Defibrillator — Defibrillation testing of cardiac defibrilator

SUMMARY:
People that have survived, or are at high risk of a lifethreatening ventricular arrhythmia are routinely offered a defibrillator (ICD). An ICD is an implanted device which can recognise a ventricular arrhythmia and then try to treat it, either by rapidly pacing the heart or by shocking the heart. Currently, very fast ventricular arrhythmias, known as VF, can only be treated with a shock. Patients find shocks painful and this study is intended to find out whether it is possible to pace the heart at very high rates during VF. It is hoped that if this is possible, further research could lead to effective treatment of VF with pacing rather than shocks, and therefore better outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years of age; Any patient with a Medtronic cardiac implantable defibrillator undergoing defibrillation testing; No contra indication to defibrillation testing Patient is able to give informed consent.

Exclusion Criteria:

* Patient is younger than 18 years; Patient is not able to give informed consent or is unwilling to participate in the study; Patient has a contraindication to defibrillation testing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
Rapid pacing of the heart | 10 seconds
  The primary outcome measure is to determine whether it is possible to obtain ventricular capture of the heart by repetitive pacing at very high rates during ventricular fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom